CLINICAL TRIAL: NCT03654326
Title: A Phase 2a, Proof of Concept, Randomized, Double-Blind, Placebo-Controlled Clinical Trial, to Evaluate the Efficacy and Safety of MK-7264 in Women With Moderate to Severe Endometriosis-Related Pain
Brief Title: A Study to Evaluate the Efficacy and Safety of Gefapixant (MK-7264) in Women With Endometriosis-Related Pain (MK-7264-034)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7264-034; MK-7264-034 (Other: MSD Protocol Number); 2018-001098-26 (EudraCT Number)
Record Dates: First submitted 2018-08-17; First posted 2018-08-31 (Actual); Results first posted 2021-07-07 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Endometriosis-related Pain
MeSH Terms: interventions — Gefapixant; Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Gefapixant (Experimental): Participants will receive a gefapixant 45 mg tablet twice a day for approximately 8 weeks (2 menstrual cycles). Naproxen sodium 275 mg tablets will also be provided to participants for use as rescue medication for endometriosis-related pain.
  Interventions: Drug: Gefapixant; Drug: Placebo; Drug: Naproxen
- Placebo (Placebo Comparator): Participants will receive a placebo matching gefapixant tablet twice a day for approximately 8 weeks (2 menstrual cycles). Naproxen sodium 275 mg tablets will also be provided to participants for use as rescue medication for endometriosis-related pain.
  Interventions: Drug: Placebo; Drug: Naproxen

INTERVENTIONS:
Drug: Gefapixant — Gefapixant tablet 45 mg taken orally
  Other Names: MK-7264
  Arms: Gefapixant
Drug: Placebo — Placebo matching gefapixant tablet taken orally
Drug: Naproxen — Naproxen sodium 275 mg tablets taken orally as needed, at dose prescribed by sites' principal investigator

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, and tolerability of gefapixant (MK-7264) in premenopausal female participants with moderate to severe endometriosis-related pain. The primary hypothesis: gefapixant is superior to placebo in reducing the average daily pelvic pain score (cyclic and non-cyclic, combined) during Treatment Cycle 2.

ELIGIBILITY:
Inclusion Criteria:

* has been surgically (laparoscopy or laparotomy) diagnosed with endometriosis.
* has cyclic AND non-cyclic, moderate to severe endometriosis-related pelvic pain (overall pelvic pain score ≥5 using a 0-10 NRS, with 0 representing no pain and 10 representing extremely severe pain).
* has had spontaneous menstrual cycles before Visit 1.
* has body mass index (BMI) between 18 kg/m^2 to 40 kg/m^2 at Visit 1.
* is not pregnant, not breastfeeding, and agrees to follow the contraceptive guidance.
* must agree to switch from her usual analgesic medication to only that which is permitted in the study.

Exclusion Criteria:

* history of hysterectomy and/or bilateral oophorectomy.
* has undiagnosed vaginal bleeding.
* has chronic, non-pelvic pain not caused by endometriosis that requires chronic analgesic.
* has a clinically significant gynecologic condition identified in the screening evaluation.
* has a history of anaphylaxis or cutaneous adverse drug reaction (with or without systemic symptoms) to sulfonamide antibiotics or other sulfonamide-containing drugs.
* has a known allergy/sensitivity or contraindication to gefapixant or its excipients.
* has an allergy/sensitivity/intolerance to naproxen sodium (rescue medication) or any contraindication to its use, or has experienced asthma, urticaria, or allergic-type reactions after taking aspirin or other nonsteroidal anti-inflammatory drugs (NSAIDs).
* has a history of endometriosis-related pain that was non-responsive to treatment with combined hormonal contraceptives (CHCs), gonadotropin-releasing hormone (GnRH) antagonists, GnRH agonists, progestins, or aromatase inhibitors.
* has a positive urine pregnancy test at any time before randomization.
* has required more than 2 weeks of continuous use of narcotics for treatment of endometriosis-related pain within 6 months of Visit 1.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 187 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (78):
- United States (30):
  - Cahaba Medical Care ( Site 0750), Birmingham, Alabama
  - Synexus US Phoenix Southeast ( Site 0729), Chandler, Arizona
  - Synexus ( Site 0734), Scottsdale, Arizona
  - Lynn Institute of the Ozarks ( Site 0720), Little Rock, Arkansas
  - California Center for Clinical Research ( Site 0741), Arcadia, California
  - Artemis Institute for Clinical Research ( Site 0716), San Diego, California
  - Alta California Medical Group ( Site 0721), Simi Valley, California
  - Thameside OBGYN Center ( Site 0747), Groton, Connecticut
  - WHUSA Fine and Gillette ( Site 0751), Hamden, Connecticut
  - Florida Fertility Institute ( Site 0737), Clearwater, Florida
  - Advanced Pharma Research ( Site 0719), Cutler Bay, Florida
  - Doral Medical Research, LLC ( Site 0706), Doral, Florida
  - KO Clinical Research, LLC ( Site 0723), Fort Lauderdale, Florida
  - Well Pharma Medical Research, Corp. ( Site 0703), Miami, Florida
  - L&C Professional Medical Research Institute ( Site 0709), Miami, Florida
  - New Horizon Research Center ( Site 0717), Miami, Florida
  - Inpatient Research Clinic, LLC ( Site 0725), Miami Lakes, Florida
  - QPS Miami Research Associates ( Site 0735), South Miami, Florida
  - Lenus Research & Medical Group Llc ( Site 0702), Sweetwater, Florida
  - Southern Clinical Research Associates ( Site 0701), Metairie, Louisiana
  - Tufts Medical Center ( Site 0742), Boston, Massachusetts
  - Carolina Women's Research and Wellness Center ( Site 0715), Durham, North Carolina
  - Palmetto Clinical Research ( Site 0707), Summerville, South Carolina
  - Chattanooga Medical Research ( Site 0743), Chattanooga, Tennessee
  - Women Partners in Health ( Site 0745), Austin, Texas
  - Corpus Christi Clinic ( Site 0744), Corpus Christi, Texas
  - HD Research Corp ( Site 0738), Houston, Texas
  - PI-Coor Clinical Research, LLC ( Site 0710), Reston, Virginia
  - Clinical Research Partners, LLC. ( Site 0704), Richmond, Virginia
  - Seattle Women's: Health, Research, Gynecology ( Site 0714), Seattle, Washington
- Australia (5):
  - Paratus Clinical Kanwal ( Site 0004), Kanwal, New South Wales
  - Royal Hospital for Women ( Site 0008), Randwick, New South Wales
  - Holdsworth House Medical Practice ( Site 0009), Sydney, New South Wales
  - Royal Adelaide Hospital ( Site 0007), Adelaide, South Australia
  - Keogh Institute for Medical Research ( Site 0002), Nedlands, Western Australia
- Chile (5):
  - Hospital San Juan de Dios de La Serena ( Site 0110), La Serena, Coquimbo Region
  - Hospital San Borja Arriaran ( Site 0103), Santiago, Santiago Metropolitan
  - Clinica Indisa [Santiago, Chile] ( Site 0101), Santiago
  - Clinica Las Condes ( Site 0109), Santiago
  - Clinica Alemana de Santiago ( Site 0107), Santiago
- New Zealand (2):
  - Southern Clinical Trials - Waitemata ( Site 0200), Auckland
  - Southern Clinical Trials Ltd ( Site 0201), Christchurch
- Poland (9):
  - Prywatna Klinika Polozniczo - Ginekologiczna ( Site 0300), Bialystok
  - Indywidualna Specjalistyczna Praktyka Lekarska Krzysztof Wilk ( Site 0316), Katowice
  - SPL Chorob Kobiecych i Połoznictwa dr L. Kobielska ( Site 0339), Katowice
  - Clinical Medical Research Sp. z o.o. ( Site 0343), Katowice
  - Osrodek Badan Klinicznych Gyncentrum ( Site 0330), Katowice
  - LIFTMED ( Site 0325), Rybnik
  - Examen Sp. z o.o. ( Site 0318), Skorzewo
  - Clinical Best Solutions ( Site 0338), Warsaw
  - Marek Elias Gabinety Ginekologiczne ( Site 0331), Wroclaw
- Puerto Rico (5):
  - Cooperativa de Facultad Medica Sanacoop ( Site 0805), Bayamón
  - Ponce Health Sciences University ( Site 0804), Ponce
  - Gynecology & Endometriosis Center LLC ( Site 0806), San Juan
  - Henry A. Rodriguez-Ginorio Private Practice ( Site 0800), San Juan
  - Genes Fertility Institute Inc. ( Site 0803), San Juan
- Russia (9):
  - Kazan State Medical University ( Site 0404), Kazan'
  - Clinical Hospital #2 of Kazan city ( Site 0406), Kazan'
  - LLC Scientific Research Medical Complex Your Health. ( Site 0405), Kazan'
  - Moscow Regional Research Institute of Tocology and Gynecolog ( Site 0411), Moscow
  - State Institution of Healthcare Moscow City Clinical Hospital 13 ( Site 0408), Moscow
  - Women clinic 22 ( Site 0400), Saint Petersburg
  - NII of Obstetrics, Gynecology and Reproductology n.a. D.O. Ott ( Site 0401), Saint Petersburg
  - Uromed LLC ( Site 0410), Smolensk
  - Siberian State Medical University ( Site 0402), Tomsk
- Spain (4):
  - Hospital Sanitas La Zarzuela ( Site 0502), Aravaca, Madrid
  - Instituto de Ciencias Medicas.ICM ( Site 0500), Alicante
  - Hospital Clinic i Provincial de Barcelona ( Site 0501), Barcelona
  - Hospital Sanitas La Moraleja ( Site 0504), Madrid
- Ukraine (9):
  - Iv-Fr Reg Perinatal center State higher Educa inst Iv-Fr Nat Med University ( Site 0910), Ivano-Frankivsk
  - Medical Center Verum ( Site 0900), Kyiv
  - GI Institute of POG of NAMS of Ukraine ( Site 0905), Kyiv
  - City Clinical Hospital No. 9 ( Site 0901), Kyiv
  - Multiprofile medical center on the base of Odessa National Medical University ( Site 0908), Odesa
  - Communal not commercial institution. Ternopil City Community Hospital 2 ( Site 0903), Ternopil
  - Communal Nonprofit Enterprize Maternity Hospital 4 ( Site 0904), Zaporizhzhya
  - Communal Institution Maternity Hospital 3 ( Site 0909), Zaporizhzhya
  - Municipal Institution Zaporizhzhya Regional Clinical Hospital ( Site 0906), Zaporizhzhya

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Arbelaez F, Joeng HK, Hussain A, Sunga S, Guan Y, Chawla A, Carmona F, Lines C, Mendizabal G. Randomized, controlled, proof-of-concept trial of gefapixant for endometriosis-related pain. Fertil Steril. 2025 Feb;123(2):280-288. doi: 10.1016/j.fertnstert.2024.09.013. Epub 2024 Sep 12. PMID 39260540

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study included a baseline menstrual cycle (approximately 4 weeks) prior to randomization to either gefapixant or placebo.
Groups:
- Gefapixant: Participants received a gefapixant 45 mg tablet twice a day for approximately 8 weeks (2 menstrual cycles). Naproxen sodium 275 mg tablets were also provided to participants, as needed, for endometriosis-related pain.
- Placebo: Participants received a placebo matching gefapixant tablet twice a day for approximately 8 weeks (2 menstrual cycles). Naproxen sodium 275 mg tablets were also provided to participants, as needed, for endometriosis-related pain.
Period: Overall Study
Arm/Group | Gefapixant | Placebo
Started | 94 | 93
Completed | 88 | 87
Not Completed | 6 | 6
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Physician Decision | 0 | 1
Not completed — Unable to adhere to study schedule | 0 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gefapixant | Placebo | Total
Number analyzed (Participants) | 94 | 93 | 187
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.5 (6.6) | 34.8 (7.3) | 34.6 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 93 | 187
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 35 | 31 | 66
  Not Hispanic or Latino | 59 | 62 | 121
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 88 | 86 | 174
  More than one race | 1 | 4 | 5
  Unknown or Not Reported | 0 | 0 | 0
Average Daily Pelvic Pain Score [Mean (Standard Deviation); unit: Scores on a scale] — Pelvic pain severity was measured using a 0-10 numeric rating scale (NRS), with 0 representing no pain and 10 representing extremely severe pain. The average of the daily pelvic pain scores entered in participants' electronic diaries (eDiaries) was calculated for the baseline cycle (approximately 28 days).
  Scores on a scale | 6.5 (1.0) | 6.5 (1.0) | 6.5 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average Daily Pelvic Pain Score During Treatment Cycle 2
Description: Pelvic pain (cyclic pain associated with menses, and non-cyclic pain not associated with menses) severity score was measured using a 0-10 numeric rating scale (NRS), with 0 representing no pain and 10 representing extremely severe pain. The averages of the daily pelvic pain scores (cyclic and non-cyclic, combined) entered in participants' electronic diaries (eDiaries) were calculated for Baseline and Treatment Cycle 2 (approximately Week 4 to Week 8). A negative change indicates a decrease in pain severity from baseline.
Time Frame: Baseline and Treatment Cycle 2 (Week 4 to Week 8; each cycle is approximately 28 days)
Population: All randomized participants who received at least one dose of double-blind study intervention and had at least one day of eDiary entries during the post-randomization treatment cycle.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a Scale
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 94 | 93
Scores on a Scale | -2.2 [-2.79 to -1.62] | -1.7 [-2.30 to -1.13]
Statistical Analysis 1: Comparison: Gefapixant vs Placebo; Test type: Superiority; p = 0.066, ANCOVA — Based on the longitudinal analysis of covariance (ANCOVA) model including factors for average pelvic pain scores at baseline cycle, stratum, treatment, cycle, interaction of stratum-by-cycle, and the interaction of treatment-by-cycle as covariates; Difference in Least Squares Mean = -0.5, 95% CI 2-sided [-1.01 to 0.03]

2. Primary Outcome: Percentage of Participants Who Experienced an Adverse Event
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. Per protocol, this analysis included AEs reported up to 14 days after end of study intervention.
Time Frame: Up to approximately 10 weeks
Population: All randomized participants who received at least one dose of study intervention.
Measure: Number; unit: Percentage of Participants
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 94 | 93
Percentage of Participants | 53.2 | 35.5
Statistical Analysis 1: Comparison: Gefapixant vs Placebo; Test type: Other — Difference in percentage of participants who experienced one or more adverse events; Difference in % vs Placebo = 17.7, 95% CI 2-sided [3.4 to 31.3] — Based on Miettinen & Nurminen method

3. Primary Outcome: Percentage of Participants Who Discontinued Study Drug Due to an Adverse Event
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Time Frame: Up to approximately 8 weeks
Population: All randomized participants who received at least one dose of study intervention.
Measure: Number; unit: Percentage of Participants
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 94 | 93
Percentage of Participants | 3.2 | 0.0
Statistical Analysis 1: Comparison: Gefapixant vs Placebo; Test type: Other — Difference in percentage of participants who discontinued study drug due to an adverse event; Difference in % vs Placebo = 3.2, 95% CI 2-sided [-0.9 to 9.0] — Based on Miettinen & Nurminen method

4. Secondary Outcome: Change From Baseline in Average Daily Cyclic Pelvic Pain Score During Treatment Cycle 2
Description: Cyclic pelvic pain (associated with menses) severity score was measured using a 0-10 NRS, with 0 representing no pain and 10 representing extremely severe pain. The average of the daily cyclic pelvic pain scores entered in participants' eDiaries was calculated for Baseline and Treatment Cycle 2 (Week 4 to Week 8). A negative change indicates a decrease in pain severity from baseline.
Time Frame: Baseline and Treatment Cycle 2 (Week 4 to Week 8; each cycle is approximately 28 days)
Population: All randomized participants who received at least one dose of double-blind study intervention, had at least one day of eDiary entry during the post-randomization treatment cycle, and had available cyclic pelvic pain score data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a Scale
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 89 | 90
Scores on a Scale | -2.0 [-2.55 to -1.35] | -1.3 [-1.94 to -0.73]
Statistical Analysis 1: Comparison: Gefapixant vs Placebo; Test type: Other — The difference in least squares mean was based on the longitudinal analysis of covariance (ANCOVA) model including factors for average pelvic pain scores at baseline cycle, stratum, treatment, cycle, interaction of stratum-by-cycle, and the interaction of treatment-by-cycle as covariates; Difference in Least Squares Mean = -0.6, 95% CI 2-sided [-1.18 to -0.06]

5. Secondary Outcome: Change From Baseline in Average Daily Non-Cyclic Pelvic Pain Score During Treatment Cycle 2
Description: Non-cyclic pelvic pain (not associated with menses) severity score was measured using a 0-10 NRS, with 0 representing no pain and 10 representing extremely severe pain. The average of the non-cyclic daily pelvic pain scores entered in participants' eDiaries was calculated for the Baseline and Treatment Cycle 2 (Week 4 to Week 8). A negative change indicates decrease in pain severity from baseline.
Time Frame: Baseline and Treatment Cycle 2 (Week 4 to Week 8; each cycle is approximately 28 days)
Population: All randomized participants who received at least one dose of double-blind study intervention, had at least one day of eDiary entry during the post-randomization treatment cycle, and had available non-cyclic pelvic pain score data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a Scale
Arm/Group | Gefapixant | Placebo
Number analyzed (Participants) | 91 | 90
Scores on a Scale | -2.3 [-2.90 to -1.69] | -1.8 [-2.40 to -1.18]
Statistical Analysis 1: Comparison: Gefapixant vs Placebo; Test type: Other — [test comment as in outcome 4, analysis 1]; Difference in Least Squares Mean = -0.5, 95% CI 2-sided [-1.04 to 0.03]

ADVERSE EVENTS:
Time Frame: All-cause mortality: Up to approximately 24 weeks Serious adverse events and other adverse events: Up to approximately 12 weeks
Description: All randomized participants who received at least one dose of study intervention
Arm/Group | Gefapixant | Placebo
All-Cause Mortality (participants affected / at risk) | 0/94 | 0/93
Serious Adverse Events (participants affected / at risk) | 0/94 | 0/93
Other Adverse Events (participants affected / at risk) | 36/94 | 12/93
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gefapixant (N=94) | Placebo (N=93)
Diarrhoea (Gastrointestinal disorders) | 6 (6) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 6 (6) | 2 (2)
Ageusia (Nervous system disorders) | 9 (9) | 1 (1)
Dysgeusia (Nervous system disorders) | 15 (16) | 2 (2)
Headache (Nervous system disorders) | 4 (4) | 7 (7)
Hypogeusia (Nervous system disorders) | 5 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-09): https://cdn.clinicaltrials.gov/large-docs/26/NCT03654326/Prot_SAP_000.pdf